CLINICAL TRIAL: NCT01325532
Title: Efficacy and Safety of Cranial Electrical Stimulation (CES) for the Treatment of Major Depressive Disorder (MDD): A Pilot Study
Brief Title: Efficacy and Safety of Cranial Electrical Stimulation (CES) for Major Depressive Disorder (MDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Fisher Wallace Labs, LLC (Unknown)
Responsible Party: Principal Investigator, David Mischoulon, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010 P000461
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; Major Depressive Disorder; MDD; Cranial Electrical Stimulation; CES
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active CES (Experimental): Active CES: The FW-100 Cranial Stimulator headset was placed on the scalp over the two dorsolateral prefrontal cortex areas. The power knob was turned to maximum setting. The waveform contains a 15000Hz square wave carrier from 0-4 mAmp. The first 15Hz modulating signal provides 50msec of "on" and 16.7msec of "off" time (total 66.7msec, 50% duty cycle). A second 500Hz modulating signal changes the "on" time series of 15000Hz pulses (750 pulses/50msec) into 25 smaller bursts of 15 pulses of the 15000Hz carrier signal, for 375 pulses in 50msec. The consecutive positive burst and "off" time is followed by an opposite negative burst and "off" time, balancing the current component to zero. Output voltage ranges from 0-40V, positive and negative. CES automatically shut off after 20 mins.
  Interventions: Device: Active CES
- Sham CES (Sham Comparator): Shame CES: The sham devices were modified to not deliver current to the headset. The current from the active device departs from the posts at the top of the device into the headsets, creating a loop when the headset is worn by the subject with the wet electrode sponges. This loop is eliminated in the sham devices by wrapping wire around the posts, thus containing the loop within the device, with no electricity leaving the headsets. This approach allows the loop to be maintained, and therefore all of the device's green and yellow amperage lights still light up, protecting the blind.
  Interventions: Device: Sham CES

INTERVENTIONS:
Device: Active CES — CES current
  Other Names: FW-100 Fisher Wallace Cranial Stimulator; Formerly known as: Liss Cranial Stimulator Model SBL202-B
  Arms: Active CES
Device: Sham CES — Sham CES (device off) for 20-minutes each day 5 days/week for 3 weeks.
  Other Names: FW-100 Fisher Wallace Cranial Stimulator (sham setting); Formerly known as: Liss Cranial Stimulator Model SBL202-B
  Arms: Sham CES

SUMMARY:
The purpose of this study is to see if using Cranial Electrical Stimulation (CES) helps improve symptoms of major depressive disorder (MDD). The investigators are studying the device's effectiveness in treating depression, as well as its safety. This is a pilot study.

Eligible participants will be randomly assigned to receive either active CES or sham CES, every weekday for 3 weeks. During the visits, subjects will receive CES or sham CES treatment for 20 minutes.

The primary outcome measure will be change in score on the HAM-D 17. The secondary outcome measure will be change in patient-reported sleep score.

DETAILED DESCRIPTION:
We examined efficacy and safety of one specific cranial electrical stimulator (CES) device at a fixed setting in subjects with treatment-resistant major depressive disorder (MDD). Thirty subjects with MDD and inadequate response to standard antidepressants were randomized to 3 weeks of treatment with CES (15/500/15000 Hz, symmetrical rectangular biphasic current of 1-4 mAmp, 40 Volts) or sham CES (device off) for 20 minutes, 5 days per week. The primary outcome measure was improvement in the 17-item Hamilton Depression Rating Scale (HAM-D-17). Adverse effects (AEs) were assessed using the Patient Related Inventory of Side Effects (PRISE). We hypothesized that subjects who received active as opposed to sham CES would have a significantly greater improvement in their depression symptoms. Due to the small sample, we could not hypothesize an effect size, but would calculate one to determine signal strength to guide the design of a larger, more rigorous study. As an exploratory aim, we also examined whether CES would benefit sleep.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to participate in the study:

1. Age 18-65 years old
2. Be in generally good health
3. Meet criteria for Major Depressive Disorder based on the DSM-IV
4. HAM-D-17 score ≥ 15, and ≤ 23

Exclusion Criteria

Subjects meeting any of the following criteria will not be allowed to participate in the study:

1. Taking any antidepressant medications (including natural products such as omega-3, St John's wort, and/or SAMe)
2. Having any unstable health conditions (unstable cardiovascular illness, cardiac arrhythmia, presence of a pacemaker, epilepsy and shock, fever, weakness and hypotension, or presence of a vagal nerve stimulator)
3. Having any electrical stimulation implants - i.e. pacemaker, deep brain stimulators (VNS, DBS), transcutaneous electrical nerve stimulator (TENS)
4. Psychotic or manic symptoms, or other evidence of a psychotic disorder; recent history of substance abuse or dependence
5. Electro Convulsive Therapy (ECT) during the last year
6. Previous course of Cranial Electrical Stimulation
7. Current active suicidal or self-injurious potential necessitating immediate treatment
8. In women, pregnancy, plans to conceive, or unwillingness to comply with birth control requirements
9. Depression-focused psychotherapy initiated within 90 days preceding enrollment or during participation in study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mischoulon, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program at Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mischoulon D, De Jong MF, Vitolo OV, Cusin C, Dording CM, Yeung AS, Durham K, Parkin SR, Fava M, Dougherty DD. Efficacy and safety of a form of cranial electrical stimulation (CES) as an add-on intervention for treatment-resistant major depressive disorder: A three week double blind pilot study. J Psychiatr Res. 2015 Nov;70:98-105. doi: 10.1016/j.jpsychires.2015.08.016. Epub 2015 Aug 29. PMID 26424428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by advertisement from our Depression Clinical and Research Program (DCRP). Informed consent was obtained per IRB guidelines. Investigators who screened subjects were our program's psychiatrists and psychologists, trained and certified in the use of appropriate diagnostic instruments such as the SCID and HAM-D.
Pre-assignment Details: Subjects who passed the screen visit returned a week later for the baseline visit. At that time, subjects received their first treatment (or sham) at the site for 20 minutes, including personal instruction of proper technique and electrode placement.
Period: Overall Study
Arm/Group | Active CES | Sham CES
Started | 17 | 13
Completed | 15 | 13
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Adults with MDD; the HAM-D score eligibility range was set to include subjects who were partial or non-responders (HAM-D 15-18) but not too severely depressed (HAMD ≤ 23), given CES's experimental nature.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CES | Sham CES | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 13 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.3) | 51.4 (11.9) | 48.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30
Hamilton Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale used here is a 17-item scale that measures severity of depression. Items are individually scored from 0-4 or from 0-2 depending on the item, and the individual scores for each item are added to comprise one score. Higher scores indicate greater severity of depression. Possible scores on the scale range from a minimum of zero (0) to a maximum of 52.
  units on a scale | 18.1 (1.5) | 18.7 (3.9) | 18.3 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale (HAM-D 17) Score From Baseline to Week 3
Description: The Hamilton Depression Rating Scale (HAM-D-17) used here is a 17-item scale that measures severity of depression. Items are individually scored from 0-4 or from 0-2 depending on the item, and the individual scores for each item are added to comprise one score. Higher scores indicate greater severity of depression. Possible scores on the scale range from a minimum of zero (0) to a maximum of 52. This section reports the improvement in depressive symptoms during the course of treatment, i.e. the change in overall score between baseline visit and week 3 visit. Change can occur in either direction (i.e. improvement or worsening). A score of greater than zero indicates a reduction of depressive symptoms (improvement), whereas a score of less than zero indicates an increase in depressive symptoms (worsening).
Time Frame: Baseline-Week 3
Population: Intent to treat sample with last observation carried forward for all randomized subject.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 17 | 13
units on a scale | 14.8 (6.3) | 13.6 (5.8)

2. Primary Outcome: Reported Side Effects Based on PRISE AE Scores
Description: This measures the emergence of different adverse (side) effects from treatment during the study. This section will describe the most commonly reported adverse effects. The section on adverse events will describe and detail the full range of AEs reported.
Time Frame: Baseline-Week 3
Population: Intent to treat sample with all subjects randomized.
Measure: Number; unit: number of subjects reporting
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 17 | 13
number of subjects reporting
  Poor concentration | 10 | 2
  Decreased energy | 6 | 2
  Fatigue | 5 | 2
  Anxiety | 5 | 4
  Flashing light/tingling | 5 | 0

3. Secondary Outcome: Change in Global Sleep Scores on the Pittsburgh Sleep Quality Index (PSQI) From Baseline to Week 3.
Description: The Pittsburgh Sleep Quality Index (PSQI) is a patient-rated instrument to assess sleep quality and quantity and its changes throughout the study. Scoring is based on 7 individual components. Each component is scored from 0-3. Higher scores indicate worse sleep. Total global sleep score ranges from zero (0) to 21. We report here the overall change in global sleep score for each treatment arm, i.e. the change in overall score between baseline visit and week 3 visit. Change can occur in either direction (i.e. improvement or worsening). A score of greater than zero indicates a reduction of sleep disturbance (improvement), whereas a score of less than zero indicates an increase in sleep disturbance (worsening).
Time Frame: Baseline-Week 3
Population: This is an intent to treat (ITT) analysis of all patients randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active CES | Sham CES
Number analyzed (Participants) | 17 | 13
units on a scale | 0.33 (2.02) | 0.77 (2.17)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: All subjects filled out the PRISE adverse effect instrument at each visit. Emergence of each side effect was assessed during the course of the study.
Arm/Group | Active CES | Sham CES
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 11/17 | 8/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CES (N=17) | Sham CES (N=13)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) — Constipation
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nausea or vomiting
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) — Palpitations
Orthostatic hypotension (Cardiac disorders) | 2 (2) | 0 (0) — Dizziness on standing
Increased perspiration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — increased sweating
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Headache
Tremors (Nervous system disorders) | 1 (1) | 0 (0) — Tremors
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Dizziness
Blurred vision (Eye disorders) | 1 (1) | 0 (0) — blurred vision
Ringing in ears (Ear and labyrinth disorders) | 1 (1) | 1 (1) — Ringing in ears
Difficulty urinating (Renal and urinary disorders) | 0 (0) | 1 (1) — Difficulty urinating
Frequent urination (Renal and urinary disorders) | 0 (0) | 1 (1) — Frequent urination
Menstrual irregularity (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Menstrual irregularity
Difficulty sleeping (General disorders) | 3 (3) | 2 (2) — Difficulty sleeping
Sleeping too much (General disorders) | 3 (3) | 1 (1) — Sleeping too much
Loss of sexual desire (Reproductive system and breast disorders) | 3 (3) | 1 (1) — Loss of sexual desire
Trouble achieving orgasm (Reproductive system and breast disorders) | 2 (2) | 0 (0) — Trouble achieving orgasm
Trouble with erections (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Trouble with erections
Anxiety (Psychiatric disorders) | 5 (5) | 4 (4) — Anxiety
Poor concentration (Psychiatric disorders) | 10 (10) | 2 (2) — Poor concentration
General malaise (Psychiatric disorders) | 5 (5) | 0 (0) — General malaise
Restlessness (Psychiatric disorders) | 3 (3) | 2 (2) — Restlessness
Fatigue (Psychiatric disorders) | 5 (5) | 2 (2) — Fatigue
Decreased energy (Psychiatric disorders) | 6 (6) | 2 (2) — Decreased energy
Flashing light and tingling sensation (Nervous system disorders) | 5 (5) | 0 (0) — Mild flashing light sensation in their peripheral vision and/or a tingling sensation in temples

LIMITATIONS AND CAVEATS:
The main limitations include a small sample and lack of an active comparator. Because CES did not separate from its sham counterpart in this sample of MDD patients, we cannot rule out that the benefit obtained from CES was due to placebo effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No